CLINICAL TRIAL: NCT03202472
Title: Pilot Trial Evaluating a Miniature Radiofrequency Tag for Localization of Non-palpable Breast Lesions for Surgery
Brief Title: Radiofrequency Identification Technology in Locating Non-palpable Breast Lesions in Patients Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-000668; NCI-2017-01097 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCLA LOCalizer 00 I; 17-000668 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-06

CONDITIONS: Breast Neoplasm; Lesion
MeSH Terms: conditions — Breast Neoplasms | interventions — Radio Frequency Identification Device; High-Energy Shock Waves

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Diagnostic (radiofrequency-guided localization) (Experimental): Patients undergo mammogram or ultrasound for image-guided placement of the radiofrequency tag within 30 days of surgery and then undergo radiofrequency-guided localization during surgery.
  Interventions: Device: Implanted Medical Device; Procedure: Mammography; Other: Questionnaire Administration; Procedure: Radiofrequency (RFID) -Guided Localization; Procedure: Ultrasonography

INTERVENTIONS:
Device: Implanted Medical Device — Radiofrequency tag
  Other Names: IMPLANTED
Procedure: Mammography — Undergo mammogram for image-guided placement of radiofrequency tag
Other: Questionnaire Administration — Ancillary studies
Procedure: Radiofrequency (RFID) -Guided Localization — Undergo radiofrequency-guided localization
  Other Names: RFID Localization; RFID-Guided Localization
Procedure: Ultrasonography — Undergo ultrasound for image-guided placement of radiofrequency tag
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; ULTRASOUND; Ultrasound Imaging; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This pilot clinical trial studies radiofrequency technology in locating non-palpable breast lesions in patients undergoing surgery. Placing a miniature radiofrequency tag or microchip in the breast lesion before surgery and using a handheld device to guide doctors during surgery may improve surgical outcomes in patients with non-palpable breast lesions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the feasibility of utilizing a new Federal Drug Administration (FDA)-cleared radiofrequency tag for localization of non-palpable breast lesions and provide preliminary data for a larger study.

OUTLINE:

Patients undergo mammogram or ultrasound for image-guided placement of the radiofrequency tag within 30 days of surgery and then undergo radiofrequency-guided localization during surgery.

After completion of study, patients are followed up within 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent to participate in the study
* Able to read and write English
* Patients with breast lesions that are non-palpable that require surgical removal
* Lesions and/or clip targetable with image guidance

Exclusion Criteria:

* Multicentric breast cancer
* Stage IV breast cancer
* Pregnant or lactating females

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maggie DiNome, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] DiNome ML, Kusske AM, Attai DJ, Fischer CP, Hoyt AC. Microchipping the breast: an effective new technology for localizing non-palpable breast lesions for surgery. Breast Cancer Res Treat. 2019 May;175(1):165-170. doi: 10.1007/s10549-019-05143-w. Epub 2019 Jan 28. PMID 30689105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: Patient consent and enrollment began 9-Aug-2017 and the final surgical procedure was performed 12-Jan-2018.
  Fifty-five patients were accessed for eligibility. Five patients who initially consented for the study but then withdrew prior to intervention because their surgeries were either cancelled or rescheduled
Pre-assignment Details: There are no pre- assignment details to describe
Groups:
- Diagnostic (Radiofrequency-guided Localization): Patients undergo mammogram or ultrasound for image-guided placement of the radiofrequency tag within 30 days of surgery and then undergo radiofrequency-guided localization during surgery.
  Implanted Medical Device: Radiofrequency tag
  Mammography: Undergo mammogram for image-guided placement of radiofrequency tag
  Questionnaire Administration: Ancillary studies
  Radiofrequency-Guided Localization: Undergo radiofrequency-guided localization
  Ultrasonography: Undergo ultrasound for image-guided placement of radiofrequency tag
Period: Overall Study
Arm/Group | Diagnostic (Radiofrequency-guided Localization)
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Radiofrequency-guided Localization)
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 60 [35 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50
Imaging Diagnosis [Count of Participants; unit: Participants]
  Mammogram | 26
  Ultrasound | 24
Lesion Diagnosis [Count of Participants; unit: Participants]
  Benign | 17
  Cancerous | 33
Lesion Category [Count of Participants; unit: Participants]
  Atypical ductal hyperplasia (ADH) | 3
  Ductal carcinoma in situ (DCIS) | 5
  DCIS with microinvasion | 1
  Encapsulated papillary carcinoma | 1
  Fibroadenoma with atypia | 1
  Glomus tumor | 1
  Invasive ductal carcinoma (IDC) | 23
  Invasive lobular carcinoma (ILC) | 3
  Lobular neoplasia | 1
  Papilloma | 3
  Phyllodes, benign | 1
  Radial Scar | 5
  Stromal Fibrosis | 2

OUTCOME MEASURES:

1. Primary Outcome: Patients With Successful Placement of the Radiofrequency Tag Under Radiographic Guidance Confirmed by Mammography
Description: Patients with successful radiofrequency tag placement
Time Frame: at time of device placement, confirmed by mammography
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Radiofrequency-guided Localization)
Number analyzed (Participants) | 50
Participants | 50

2. Primary Outcome: Patients With Successful Retrieval of the Radiofrequency Tag Confirmed by Specimen Radiography
Description: Patients with successful radiofrequency tag retrieval.
Time Frame: at time of surgery, within 30 days of tag implant
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Radiofrequency-guided Localization)
Number analyzed (Participants) | 50
Participants | 50

3. Secondary Outcome: Days Prior to Surgery of Insertion of Marker
Description: Mean number of days before surgery that radiofrequency tag was placed.
Time Frame: Up to 30 days prior to surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Diagnostic (Radiofrequency-guided Localization)
Number analyzed (Participants) | 50
days | 1.4 (2.8)

4. Secondary Outcome: Patient Experience With Image-guided Placement of Tag as Rated by a Patient Questionnaire
Description: The patient experience with image-guided placement of the radio frequency Identification (RFID) tag.This assessments was captured using Likert-type questionnaires. Individual question responses for the patient and physician questionnaires ranged from 1 to 5 with the score of 5 representing the maximum positive or favorable response to each question. The following choices were included in each questionnaire:
  1. Strongly disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
  Responses of the individual scales were added to create a total score, which would include a possible total range of 5 to a maximum of 25 points. 25 is the maximum positive or favorable response.
Time Frame: within 24 hours of device placement
Population: All Patients
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diagnostic (Radiofrequency-guided Localization)
Number analyzed (Participants) | 50
units on a scale | 21.3 (3.9)

5. Secondary Outcome: Patients With Cancer Requiring Re-excision
Description: Patients requiring re-excision.
Time Frame: up to 4 weeks post initial surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Radiofrequency-guided Localization)
Number analyzed (Participants) | 50
Participants | 2

6. Secondary Outcome: Patients With Documented Migration of Marker
Description: Movement of radiofrequency tag from point of placement
Time Frame: at time of surgery, within 30 days of tag implant
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Radiofrequency-guided Localization)
Number analyzed (Participants) | 50
Participants | 0

7. Secondary Outcome: Patients With Positive Margins on Initial Lumpectomy Using Radiofrequency Identification Technology
Description: Patients with margins of excisable tissue remaining.
Time Frame: at time of pathologic evaluation of surgical specimen, within 4 weeks of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (Radiofrequency-guided Localization)
Number analyzed (Participants) | 50
Participants | 4

8. Secondary Outcome: Radiologist's Experience Placing Radiofrequency Tag Compared to Wire Localization as Measured by a Radiologist's Questionnaire
Description: The radiologist's experience with image-guided placement of the RFID tag.This assessments was captured using Likert-type questionnaires. Individual question responses for the patient and physician questionnaires ranged from 1 to 5 with the score of 5 representing the maximum positive or favorable response to each question. The following choices were included in each questionnaire:
  1. Strongly disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
  Responses of the individual scales were added to create a total score, which would include a possible total range of 5 to a maximum of 25 points. 25 is the maximum positive or favorable response.
Time Frame: within 24 hours of device placement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diagnostic (Radiofrequency-guided Localization)
Number analyzed (Participants) | 50
units on a scale | 20.4 (2.4)

9. Secondary Outcome: Surgeon's Experience Using Radiofrequency Tag to Guide Resection Compared to Wire Localization as Measured by a Surgeon's Questionnaire
Description: The surgeon's experience with image-guided placement of the RFID tag.This assessments was captured using Likert-type questionnaires. Individual question responses for the patient and physician questionnaires ranged from 1 to 5 with the score of 5 representing the maximum positive or favorable response to each question. The following choices were included in each questionnaire:
  1. Strongly disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
  Responses of the individual scales were added to create a total score, which would include a possible total range of 5 to a maximum of 25 points. 25 is the maximum positive or favorable response.
Time Frame: within 24 hours of surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diagnostic (Radiofrequency-guided Localization)
Number analyzed (Participants) | 50
units on a scale | 21.5 (2.7)

10. Secondary Outcome: Volume (cm3), of Tissue Removed With Specimen With Tag (Not Including Shave Margins, if Taken)
Description: Amount of tissue removed with radiofrequency tag.
Time Frame: at time of pathologic evaluation of surgical specimen, within 4 weeks of surgery
Measure: Mean (Standard Deviation); unit: CM3
Arm/Group | Diagnostic (Radiofrequency-guided Localization)
Number analyzed (Participants) | 50
CM3 | 30.7 (26.4)

ADVERSE EVENTS:
Time Frame: Adverse event reports were completed routinely for the first 20 patients enrolled in the study within 24 hours of device placement. Final monitoring for adverse events was performed at the time of the post-operative visit, which occurred within 14 days of surgery. The final monitoring occurred for the last patient on 01/23/2018
Arm/Group | Diagnostic (Radiofrequency-guided Localization)
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT03202472/Prot_SAP_000.pdf
  • Informed Consent Form (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT03202472/ICF_002.pdf